CLINICAL TRIAL: NCT02100475
Title: A Trial Comparing Sequential Addition of Insulin Aspart Versus Further Dose Increase With Insulin Degludec/Liraglutide in Subjects With Type 2 Diabetes Mellitus, Previously Treated With Insulin Degludec/Liraglutide and Metformin and in Need of Further Intensification (DUAL™ - Intensification)
Brief Title: A Trial Comparing Sequential Addition of Insulin Aspart Versus Further Dose Increase With Insulin Degludec/Liraglutide in Subjects With Type 2 Diabetes Mellitus, Previously Treated With Insulin Degludec/Liraglutide and Metformin and in Need of Further Intensification
Acronym: DUAL™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4119; 2013-002878-47 (EudraCT Number); U1111-1145-0183 (Other: WHO)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide + Metformin (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Insulin degludec/liraglutide + Insulin Aspart + Metformin (Active Comparator)
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Insulin degludec/liraglutide will be given subcutaneously (s.c., under the skin) once daily in combination with metformin.
  Dose individually adjusted.
Drug: insulin aspart — Dose titration of insulin aspart will be based on the respective pre-meal(s) and bedtime SMPG measured daily.
  Arms: Insulin degludec/liraglutide + Insulin Aspart + Metformin

SUMMARY:
This trial is conducted globally. The aim of the trial is to compare sequential addition of insulin aspart versus further dose increase with insulin degludec/liraglutide in subjects with type 2 diabetes mellitus, previously treated with insulin degludec/liraglutide and metformin and in need of further intensification.

This is an extension to trial NN9068-3952, NCT01952145 (DUAL™ V).

ELIGIBILITY:
Inclusion Criteria:

* Completion (Visit 28) of NN9068-3952 with insulin degludec/liraglutide + metformin
* HbA1c (glycosylated haemoglobin) above or equal to 7 percent at Visit 27 of NN9068-3952 trial

Exclusion Criteria:

* Clinically significant diseases of the major organ systems
* Screening calcitonin above or equal to 50 ng/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (54):
- United States (7):
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Renton, Washington
- Argentina (5):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Corrientes
  - Novo Nordisk Investigational Site, Salta
  - Novo Nordisk Investigational Site, Zárate
- Australia (5):
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, Herston, Queensland
  - Novo Nordisk Investigational Site, Ipswich, Queensland
  - Novo Nordisk Investigational Site, Robina, Queensland
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
- Greece (4):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Ioannina
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (4):
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Győr
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Miskolc
- Mexico (4):
  - Novo Nordisk Investigational Site, Pachuca, Hidalgo
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Monterrey
- Russia (7):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Kirov
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Volgograd
- Slovakia (9):
  - Novo Nordisk Investigational Site, Bardejov
  - Novo Nordisk Investigational Site, Dolný Kubín
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Poprad
  - Novo Nordisk Investigational Site, Považská Bystrica
  - Novo Nordisk Investigational Site, Prievidza
  - Novo Nordisk Investigational Site, Trnava
  - Novo Nordisk Investigational Site, Veľký Meder
- South Africa (4):
  - Novo Nordisk Investigational Site, Midrand, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Alberton
- Spain (5):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 19 sites in 8 countries as follows: Argentina: 2 sites; Greece: 2 sites, Hungary: 1 site; Russian Federation: 5 sites; Slovakia: 4 sites, South Africa: 1 site; Spain: 1 site, United States: 3 sites.
Pre-assignment Details: Subjects with type 2 diabetes mellitus who were inadequately controlled (HbA1c level ≥ 7% [53 mmol/mol]) on treatment with IDegLira and metformin after 26 weeks of treatment in the NN9068-3952 trial were screened. Eligible subjects were randomised in a 1:1 manner to one of the two parallel treatment groups (IDegLira or IDegLira + IAsp).
Groups:
- IDegLira: Insulin degludec/liraglutide (IDegLira) was given subcutaneously (s.c., under the skin) once daily in combination with metformin. The starting dose of IDegLira was the dose of IDegLira used at the end of the NN9068-3952 trial. Intensification with IDegLira was performed by dose optimisation up to a maximum of 80 dose steps (80 units IDeg/2.9 mg Lira). All subjects continued with metformin at pre-trial doses (≥ 1500 mg or the maximum tolerated dose).
- IDegLira + IAsp: IDegLira was given subcutaneously (s.c., under the skin) once daily in combination with metformin. The starting dose of IDegLira was the dose of IDegLira used at the end of the NN9068-3952 trial. IDegLira was titrated up to a maximum dose of 50 dose steps (50 units IDeg/1.8 mg Lira) with sequential add-on of bolus insulin aspart (IAsp). Dose titration of insulin aspart was based on the respective premeal(s) and bedtime self-measured plasma glucose (SMPG) measured daily. All subjects continued with metformin at pre-trial doses (≥ 1500 mg or the maximum tolerated dose).
Period: Overall Study
Arm/Group | IDegLira | IDegLira + IAsp
Started | 16 | 15
Completed | 14 | 13
Not Completed | 2 | 2
Not completed — Unclassified | 1 | 2
Not completed — Withdrawal criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for full analysis set (FAS = 31 subjects).
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegLira | IDegLira + IAsp | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (11.7) | 57.4 (11.2) | 57.4 (11.3)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 7 | 7 | 14
HbA1c [Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin] | 7.6 (0.9) | 7.7 (0.7) | 7.6 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: Full analysis set (FAS) included all randomised subjects (31 subjects). Missing data were imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | IDegLira | IDegLira + IAsp
Number analyzed (Participants) | 16 | 15
Percentage of glycosylated haemoglobin | -0.43 (0.94) | -0.14 (1.09)
Statistical Analysis 1: Comparison: IDegLira vs IDegLira + IAsp; The response and change from baseline in the response after 26 weeks of treatment was analysed using an analysis of covariance (ANCOVA) method with treatment and baseline IDegLira dose strata as fixed factors and baseline response as a covariate. Missing data were imputed using LOCF; Test type: Superiority or Other; p = 0.427, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.05 to 0.46]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: FAS included all randomised subject (31 subjects). Missing data were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | IDegLira | IDegLira + IAsp
Number analyzed (Participants) | 16 | 15
Kilograms | 0.9 (2.1) | 1.5 (3.2)

3. Secondary Outcome: Number of Treatment-emergent Confirmed Hypoglycaemic Episodes
Description: Treatment-emergent hypoglycaemic episodes: if the onset of the episode occurred on or after the first day of investigational medicinal product administration, and no later than 7 days after the last day on investigational medicinal product. Confirmed hypoglycaemia: subject unable to treat himself/herself and/or have a recorded plasma glucose < 3.1 mmol/L (56 mg/dL).
Time Frame: Week 0 - 26
Population: Safety analysis set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (31 subjects). Confirmed hypoglycaemic episodes were reported by 2 subjects in IDegLira arm and 2 subjects in IDegLira + IAsp arm.
Measure: Number; unit: Number of episodes
Arm/Group | IDegLira | IDegLira + IAsp
Number analyzed (Participants) | 16 | 15
Number of episodes | 34 | 4

ADVERSE EVENTS:
Time Frame: From first trial-related activity (week 0) after the subject had signed the informed consent until the end of the post-treatment follow-up period (week 27).
Description: SAS included all subjects receiving at least one dose of the investigational product or comparator, (SAS = 31 subjects).
  A treatment-emergent adverse event (TEAE) was defined as an event that had an onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment.
Arm/Group | IDegLira | IDegLira + IAsp
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/15
Other Adverse Events (participants affected / at risk) | 11/16 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=16) | IDegLira + IAsp (N=15)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=16) | IDegLira + IAsp (N=15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the small number of subjects in this trial, the data should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of trial, one or more scientific publications may be prepared collaboratively by the investigators and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.